CLINICAL TRIAL: NCT04150094
Title: Intravaginal Vibratory Stimulus and Pelvic Floor Muscle Training to Treat Female Urinary Incontinence: a Randomized Clinical Trial
Brief Title: Intravaginal Vibratory Stimulus and Pelvic Floor Muscle Training
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the covid pandemic.
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0354
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor muscle training (PFMT) (Active Comparator): Pelvic floor muscle training without stimulus.
  Interventions: Other: Pelvic floor muscle training (PFMT)
- Pelvic floor muscle training + intravaginal vibratory stimulus (Experimental): Pelvic floor muscle training with intravaginal vibratory stimulation.
  Interventions: Other: Pelvic floor muscle training + intravaginal vibratory stimulus

INTERVENTIONS:
Other: Pelvic floor muscle training (PFMT) — Participants will be firstly evaluated and orientated about pelvic floor muscles and pelvic floor muscle training. They will be clarified about the role of pelvic floor muscles in continence mechanisms and will be orientated to perform 8 weeks of PFMT without stimulus, coming once a week to a session supervised by physiotherapist and will be encouraged to perform the exercises at home during the other week days.
  Arms: Pelvic floor muscle training (PFMT)
Other: Pelvic floor muscle training + intravaginal vibratory stimulus — Participants will be firstly evaluated and orientated about pelvic floor muscles and pelvic floor muscle training. They will be clarified about the role of pelvic floor muscles in continence mechanisms and will be orientated to perform 8 weeks of PFMT with intravaginal vibratory stimulus. They will need to come once a week to a session supervised by physiotherapist to use the vibration device and will be encouraged to perform the exercises at home during the other week days.
  Arms: Pelvic floor muscle training + intravaginal vibratory stimulus

SUMMARY:
This is a randomized blinded trial with non-probabilistic sampling for convenience. Our goal is to compare PFMT with intravaginal vibratory stimulus versus PFMT alone on the treatment of female urinary incontinence.

DETAILED DESCRIPTION:
This is a randomized blinded trial with non-probabilistic sampling for convenience. Our goal is to compare PFMT with intravaginal vibratory stimulus versus PFMT alone on the treatment of female urinary incontinence. Women with an indication for conservative treatment of urinary incontinence will be referred to the Pelvic Floor Physiotherapy Team by the Medical Team of the Ambulatory of Urogynecology and Obstetrics of the Hospital de Clínicas de Porto Alegre and those who are in compliance with the inclusion criteria proposed for the research will be invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women with urinary incontinence;
* Know how to perform a voluntary pelvic floor muscle contraction;
* Have not undergone pelvic floor muscle training in the last 6 months;
* Understand the instruments used in research.

Exclusion Criteria:

* Latex allergy;
* Neurological diseases;
* Pelvic organ prolapse > grade 2;
* Pain during vaginal palpation and / or introduction of the vaginal probe;
* Vaginal atrophy;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in urinary incontinence | 8 weeks
  We will measure it using the "International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) - Portuguese version", pre and post treatment, to assess if there are any changes in bladder control after the protocols. It consists of 3 scored items which evaluate the frequency, volume of leakage and overall impact of incontinence. The overall score ranges from 0 to 21, with greater values indicating increased severity. Klovning et al (2009) says that ICIQ-SF may be divided into the following four severity categories of UI: slight (1-5), moderate (6-12), severe (13-18) and very severe (19-21). Lim et al (2019) suggested that for women undergoing nonsurgical treatments for incontinence, reductions of 4 points in ICIQ-UI SF are perceived as clinically meaningful.

SECONDARY OUTCOMES:
Impact in quality of life | 8 weeks
  We are using the "International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) - Portuguese version", which asks about overall impact of UI in quality of life by a scale from 0-10 of how much these symptoms bothered the patient's life. We are going to say the participant "imagine that 0 is if urinary leakage doesn't bother you at all and 10 is as much as this can disrupt your life". There are other questions in this questionnaire according to the severity of the UI symptoms. Each answer has a punctuation and the total score could range between 0 and 21. The higher, the worse is the severity of UI and the impact on the participant's quality of life. The ICIQ is highly recommended (Grade A) for the basic evaluation of the patient's perspective of urinary incontinence (Abrams et al, 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Geraldo Lopes Ramos, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- José Geraldo Lopes Ramos, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The SPSS spreadsheet with relevant research data (characterization of the sample and severity of UI) and statistical analysis may be shared by e-mail request.